CLINICAL TRIAL: NCT02353351
Title: Closure of Atrial Septal Defects With the AMPLATZER™ Septal Occluder (ASO) Post Market Surveillance Study
Brief Title: ADVANCE ASO AMPLATZER™ Atrial Septal Occluder Post Market Surveillance Study
Acronym: ASO 522
Status: Terminated | Type: Observational
Why Stopped: The sponsor's study closure justification addressed the 522 Order's questions.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: PS130046
Record Dates: First submitted 2014-12-02; First posted 2015-02-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Atrial Septal Defect Secundum
MeSH Terms: conditions — Foramen Ovale, Patent | interventions — Septal Occluder Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: atrial septal occluder — Single arm atrial septal defect closure with the AMPLATZER Septal Occluder
  Other Names: AMPLATZER Septal Occluder

SUMMARY:
Prospective, multicenter, case-cohort study.To identify potential risk factors associated with the occurrence of erosion due to implantation of the AMPLATZER™ Septal Occluder (ASO.)

DETAILED DESCRIPTION:
This study will enroll 8000 subjects. The sub-cohort will consist of 160 (2%) subjects, randomly selected from the full cohort. The analysis population will consist of all subjects in the sub-cohort, combined with all subjects with erosion events who are not in the sub-cohort. A detailed assessment of risk factors will be conducted on the subjects in this analysis population.

ELIGIBILITY:
Inclusion Criteria:

To participate in this clinical investigation, the patient must meet all of the following inclusion criteria:

1. Patient indicated for ASD closure who has echocardiographic evidence of ostium secundum atrial septal defect and clinical evidence of right ventricular volume overload (such as, 1.5:1 degree of left-to-right shunt or RV enlargement) and is implanted with the ASO device Note: This does not include the indication for closure of a fenestration following a fenestrated Fontan procedure
2. Patient is willing and able to complete the follow-up requirements of this study
3. Patient signs the informed consent (or a legal representative signs the informed consent.)

Exclusion Criteria:

Patient is not eligible for clinical investigation participation if he/she meets any of the following exclusion criteria:

1. Patient is known to have extensive congenital cardiac anomaly which can only be adequately repaired by way of cardiac surgery
2. Patient is known to have sepsis within 1 month prior to implantation, or any systemic infection that cannot be successfully treated prior to device placement
3. Patient is known to have a bleeding disorder, untreated ulcer, or any other contraindications to aspirin therapy (unless another anti-platelet agent can be administered for 6 months)
4. Patient is known to have a demonstrated intracardiac thrombus on echocardiography
5. Patient whose size (such as, too small for transesophageal echocardiography probe, catheter size) or condition (active infection, etc.) would cause the patient to be a poor candidate for cardiac catheterization
6. Patient has margins of defect that are less than 5 mm to the coronary sinus, AV valves or right upper lobe pulmonary vein

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients indicated for ASD closure have echocardiographic evidence of ostium secundum atrial septal defect and clinical evidence of right ventricular volume overload (such as, 1.5:1 degree of left-to-right shunt or RV enlargement).
  The subject population includes vulnerable patients.
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of cardiac erosion | 1 year
  Cumulative incidence of erosion will be reported as:
  • The number of erosions per 8000 subjects.

SECONDARY OUTCOMES:
Aortic Rim Measurements (< 5 mm, ≥ 5 mm) | 1 year
Atrio-Ventricular (AV) Valve Rim Measurements (< 5 mm, ≥ 5 mm) | 1 year
Superior Vena Cava (SVC) Rim Measurements (< 5 mm, ≥ 5 mm) | 1 year
Inferior Vena Cava (IVC) Rim Measurements (< 5 mm, ≥ 5 mm) | 1 year
Other Evaluable Rim Measurements (< 5 mm, ≥ 5 mm) | 1 year
Ratio of Defect Size (Diameter) to Septal Length (< 0.5:1, ≥ 0.5:1) | 1 year
Ratio of Defect Size (Diameter) to Septal Width (< 0.5:1, ≥ 0.5:1) | 1 year
Device Splaying the Aorta (Yes, No) | 1 year
Device Impingement of the Aorta (Yes, No) | 1 year
Device Abutting the Aorta (Yes, No) | 1 year
Age (< 14, ≥ 14 years) | 1 year
Gender (Male, Female) | 1 year
Device Size Implanted (< 18 mm, ≥ 18 mm) | 1 year
Device Size to Defect Size (< 1.5:1, ≥ 1.5:1) | 1 year
Body Surface Area (<1.5 m2 and ≥ 1.5m2) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Oza, Study Director — Abbott Medical Devices
Locations (65):
- United States (65):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Stanford University Medical Center, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Rady Children's Hospital, San Diego, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Iowa Heart Center / Mercy Medical Center, West Des Moines, Iowa
  - Children's Hospital, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Children's Hospital, St Louis, Missouri
  - Sunrise Hospital, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - New York Presbyterian/Cornell, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Children's Hospital of New York - Presbyterian, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - North Austin Medical Center, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Houston Methodist DeBakey Heart and Vascular Center, Houston, Texas
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston/Memorial Hermann Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Medical Research Group, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin